CLINICAL TRIAL: NCT00897104
Title: A Randomized, Placebo-Controlled, Parallel-Groups, Outpatient Study to Compare the Efficacy and Safety of MK0462 5 mg p.o. and Sumatriptan 50 mg p.o. for the Acute Treatment of Migraine
Brief Title: MK0462 5 mg, Sumatriptan 50 mg, and Placebo Comparison Study (0462-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-029; 2009_593
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): Rizatriptan
  Interventions: Drug: rizatriptan benzoate (MK0462)
- 2 (Experimental): Sumatriptan
  Interventions: Drug: Comparator: sumatriptan
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: rizatriptan benzoate (MK0462) — single dose 5 mg rizatriptan p.o.
  Other Names: MK0462
  Arms: 1
Drug: Comparator: sumatriptan — single dose 50 mg sumatriptan p.o.
  Arms: 2
Drug: Comparator: Placebo — Placebo to rizatriptan or sumatriptan, single dose placebo tablet taken orally
  Arms: 3

SUMMARY:
A study to compare rizatriptan (MK0462) 5 mg by mouth (p.o.) and sumatriptan 50 mg p.o. for the acute treatment of a migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Participant had at least a 6-month history of migraine, with or without aura
* Participant was male, or if female, must have been postmenopausal, surgically sterilized, or taking adequate contraceptive precautions
* Participant was judged to be in good health, apart from migraine

Exclusion Criteria:

* Participant was Pregnant or a nursing mother
* Participant had a history or current evidence of drug or alcohol abuse
* Participant had a history or clinical evidence of cardiovascular disease
* Participant had a clinically significant Electrocardiography (ECG) abnormality
* Participant had a resting systolic blood pressure of greater than 145 mm Hg or diastolic of less than 95 mm Hg at screening
* Participant had received treatment with an investigational device or compound within 30 days of the study
* Participant typically suffered from less then 1 or more than 8 attacks of migraine per month
* Participant had difficulty in distinguishing his/her migraine attacks from tension or interval headaches
* Participant was currently taking monoamine oxidase inhibitors, methysergide or lithium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 933 (Actual)
Dates: Start 1995-08; Primary Completion 1996-05 (Actual); Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Ho TW, Fan X, Rodgers A, Lines CR, Winner P, Shapiro RE. Age effects on placebo response rates in clinical trials of acute agents for migraine: pooled analysis of rizatriptan trials in adults. Cephalalgia. 2009 Jul;29(7):711-8. doi: 10.1111/j.1468-2982.2008.01788.x. Epub 2009 Feb 3. PMID 19210513
- [Result] Ferrari MD, Loder E, McCarroll KA, Lines CR. Meta-analysis of rizatriptan efficacy in randomized controlled clinical trials. Cephalalgia. 2001 Mar;21(2):129-36. doi: 10.1046/j.1468-2982.2001.00169.x. PMID 11422095
- [Result] Block GA, Goldstein J, Polis A, Reines SA, Smith ME. Efficacy and safety of rizatriptan versus standard care during long-term treatment for migraine. Rizatriptan Multicenter Study Groups. Headache. 1998 Nov-Dec;38(10):764-71. doi: 10.1046/j.1526-4610.1998.3810764.x. PMID 11284464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 31 sites: 6 in UK, 9 in Norway, 2 in Switzerland, and 14 in Sweden
  First Participant Treated: August 1995
  Last Participant Treated: May 1996.
Pre-assignment Details: Participants screened at a pretreatment visit were given allocated drug supply with instructions. If participants had not treated an attack within 2 months of being enrolled, they were required to return for a rescreen visit. If by 4 months after being enrolled participants still had not treated an attack, they were discontinued from the study.
Groups:
- Rizatriptan 5 mg: Rizatriptan 5 mg orally once for treatment of single migraine attack
- Sumatriptan 5 mg: Sumatriptan 5 mg orally once for treatment of single migraine attack
- Placebo: Placebo matching Rizatriptan 5 mg or Sumatriptan 5 mg orally once for treatment of single migraine attack
Period: Overall Study
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Started | 418 (Participants who were allocated study drug) | 428 (Participants who were allocated study drug) | 87 (Participants who were allocated study drug)
Participants Treated | 355 (Participants who took study drug) | 357 (Participants who took study drug) | 80 (Participants who took study drug)
Participants Not Treated | 63 (Participants who did not take study drug) | 71 (Participants who did not take study drug) | 7 (Participants who did not take study drug)
Completed | 354 (Participants who took study drug and completed the study) | 357 (Participants who took study drug and completed the study) | 79 (Participants who took study drug and completed the study)
Not Completed | 64 | 71 | 8
Not completed — Lost to Follow-up | 12 | 17 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 23 | 27 | 3
Not completed — Abnormal Prestudy Labs | 2 | 0 | 0
Not completed — Abnormal Baseline ECG | 2 | 2 | 0
Not completed — Need for Concom. Med. | 0 | 1 | 1
Not completed — Lack of Migraine Attack | 20 | 22 | 1
Not completed — No Longer Met Inc/Exc Criteria | 1 | 0 | 0
Not completed — Other | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo | Total
Number analyzed (Participants) | 355 | 357 | 80 | 792
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.3) | 41.8 (10.1) | 44.3 (10.5) | 41.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 291 | 70 | 652
  Male | 64 | 66 | 10 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 352 | 356 | 80 | 788
  Asian | 3 | 1 | 0 | 4
Baseline Headache Severity [Number; unit: Participants] — Each participant rated headache severity on a 4-grade scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain).
  Participants
    Grades 0,1: no pain, Mild, or missing | 6 | 8 | 0 | 14
    Grade 2: Moderate | 216 | 221 | 51 | 488
    Grade 3: Severe | 133 | 128 | 29 | 290

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours After Treatment
Description: Participants reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe pain) at baseline to grades 0 or 1 (no headache or mild pain) at 2 hours after treatment
Time Frame: 2 hours after treatment
Population: An "all-participants-treated" approach was used in the primary analysis, including all participants who had at least one assessment of pain severity within 2 hours after dose. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 352 | 356 | 80
Participants
  2-hour pain relief | 223 | 238 | 18
  No 2-hour pain relief | 129 | 118 | 62

2. Primary Outcome: Time to Relief Within 2 Hours After Treatment
Description: Participants reporting time to relief (defined as the first time that a participant reported grade 0 or 1 in headache severity within 2 hours after treatment (for the comparison of rizatriptan 5 mg and sumatriptan 50 mg).
Time Frame: within 2 hours after treatment
Population: An "all-participants-treated" approach was used in the primary analysis, including all participants who had at least one assessment of pain severity within 2 hours after test medication.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 352 | 356 | 80
Participants
  First pain relief within 2 hrs | 231 | 247 | 24
  Pain relief did not occur within 2 hrs | 121 | 109 | 56

3. Secondary Outcome: Pain Free at 2 Hours After Treatment
Description: Participants pain free (defined as a reduction of headache severity to grade 0 [no pain]) at 2 hours after treatment. Each participant rated headache severity on a 4-grade scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain).
Time Frame: 2 hours after treatment
Population: An "all-participants-treated" approach was used in the secondary analysis, including all participants who had at least one assessment of pain severity within 2 hours after test medication. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 352 | 356 | 80
Participants
  2-hour pain freedom | 95 | 113 | 2
  No 2-hour pain freedom | 257 | 243 | 78

4. Secondary Outcome: Lack of Functional Disability at 2 Hours After Treatment as Measured by the Level of Impairment in Daily Activities
Description: Participants with no functional disability measured by the level of impairment to daily activities at 2 hours after treatment. Each participant rated functional disability on a 4-grade scale (0 =normal; 1 = daily activities mildly impaired; 2 = daily activities severely impaired; 3 =unable to carry out daily activities, required bed rest).
Time Frame: 2 hours after treatment
Population: An "all-participants-treated" approach was used in the secondary analysis. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 350 | 355 | 80
Participants
  Normal | 108 | 116 | 4
  Mildly Impaired | 152 | 148 | 28
  Severely Impaired | 38 | 42 | 18
  Required Bed Rest | 52 | 49 | 30

5. Secondary Outcome: Presence or Absence of Associated Symptoms (Photophobia, Phonophobia, Nausea, and Vomiting) at 2 Hours After Treatment
Description: Participants who recorded the presence or absence of the associated symptoms photophobia, phonophobia, nausea, and vomiting at 2 hours after treatment.
Time Frame: 2 hours after treatment
Population: "All-participants-treated" approach was used. Missing data were replaced by carrying forward the preceding value. Participants Analyzed For Nausea: Rizatriptan 348; Sumatriptan 352; Placebo 78. Participants Analyzed for Vomiting: Rizatriptan 342; Sumatriptan 342; Placebo 73. Number of participants analyzed is correct for the other categories.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 350 | 354 | 80
Participants
  2-hour Photophobia | 161 | 153 | 66
  No 2-hour Photophobia | 189 | 201 | 14
  2-hour Phonophobia | 126 | 125 | 47
  No 2-hour Phonophobia | 224 | 229 | 33
  2-hour Nausea | 105 | 131 | 48
  No 2-hour Nausea | 243 | 221 | 30
  Not Analyzed for Nausea | 2 | 2 | 2
  2-hour Vomiting | 12 | 12 | 6
  No 2-hour Vomiting | 330 | 330 | 67
  Not Analyzed for Vomiting | 8 | 12 | 7

6. Secondary Outcome: Participants Who Used Escape Medication 2 Hours After the Treatment Dose
Description: Escape medication is defined as rescue medication for participants who experienced lack of efficacy from the study medication.
Time Frame: 2 hours after treatment
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 355 | 357 | 80
Participants
  Used Escape Medication | 73 | 55 | 33
  Did not Use Escape Medication | 282 | 302 | 47

7. Secondary Outcome: Duration of Relief (Time to Recurrence From the Time of First Recorded Pain Relief [Grade = 0 or 1])
Description: Duration of relief or the time to recurrence from the time of first recorded pain relief (grade = 0 or 1) was calculated for responders who had a headache recurrence
Time Frame: 24 hours
Population: The duration of relief, or the time to recurrence from the time of first recorded pain relief (grade = 0 or 1), was calculated for responders who had a headache recurrence.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Number analyzed (Participants) | 84 | 80 | 6
Hours | 11.07 (6.56) | 11.58 (5.86) | 14.38 (5.00)

ADVERSE EVENTS:
Time Frame: During the 24 hours treatment period, and up to and including 7 days after the last dose of study therapy.
Description: Although a participant may have had two or more adverse experiences the participant is counted only once in a category. The same participant may appear in different categories.
  The At Risk population are the participants that received study treatment.
Arm/Group | Rizatriptan 5 mg | Sumatriptan 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/355 | 0/357 | 0/80
Other Adverse Events (participants affected / at risk) | 92/355 | 108/357 | 16/80
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=355) | Sumatriptan 5 mg (N=357) | Placebo (N=80)
Asthenia/Fatigue (General disorders) | 25 | 18 | 1
Fever (General disorders) | 1 | 1 | 1
Pain, Abdominal (General disorders) | 4 | 5 | 0
Pain, Chest (General disorders) | 8 | 16 | 0
Warm Sensation (General disorders) | 4 | 3 | 1
Palpitation (Cardiac disorders) | 2 | 6 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 10 | 9 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 13 | 21 | 2
Pain, Mouth (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0
Heaviness, Regional (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Pain, Back (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Pain, Neck (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2
Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0
Strain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Apathy (Psychiatric disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 13 | 17 | 4
Dream Abnormality (Psychiatric disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 7 | 6 | 0
Hypesthesia (Nervous system disorders) | 4 | 6 | 3
Mental Acuity Decreased (Nervous system disorders) | 3 | 5 | 1
Paresthesia (Nervous system disorders) | 11 | 12 | 2
Somnolence (Psychiatric disorders) | 13 | 17 | 0
Vertigo (Nervous system disorders) | 6 | 3 | 1
Discomfort, Pharyngeal (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1

LIMITATIONS AND CAVEATS:
No limitations were encountered in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.